CLINICAL TRIAL: NCT03370484
Title: The Effect of Calcium Ingestion on Gut Hormone Secretion.
Brief Title: Calcium and Gut Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Javier Gonzalez, Associate Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: REACH EP 16/17_164C
Record Dates: First submitted 2017-12-06; First posted 2017-12-12 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Water with artificial sweetener
  Interventions: Dietary Supplement: Control
- Milk mineral supplement (Experimental): Milk Minerals containing 1000 mg calcium with artificial sweetener and water
  Interventions: Dietary Supplement: Milk mineral supplement

INTERVENTIONS:
Dietary Supplement: Control — Water with 80 mg sucralose
  Arms: Control
Dietary Supplement: Milk mineral supplement — Water with milk mineral supplement (1000 mg calcium), plus 80 mg sucralose
  Arms: Milk mineral supplement

SUMMARY:
Gut hormones have therapeutic potential in the prevention and treatment obesity and type 2 diabetes (T2D). Rodent evidence suggests that calcium may stimulate gut hormone secretion. Evidence in humans however, is lacking. This study aims to assess whether the calcium ingestion stimulates gut hormone availability in humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age between 18-65 yrs.
* Able to consume provided supplement.
* Weight stable for the past 3 month (no change within 3%)

Exclusion Criteria:

* Any previous or current metabolic, cardio-pulmonary or musculoskeletal disease
* Not between the ages of 18-65 years
* A body mass index below 18.5 kg/m2 or above 30 kg/m2 (body mass (kg) divided by your height (m) squared)
* Taking medications that may influence your metabolism
* Plans to change your lifestyle (diet and/or physical activity) during the study period
* Not willing to refrain from alcohol containing drinks or unaccustomed exercise one day before the laboratory sessions.
* Current smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Postprandial plasma GLP-1 area under the curve (mmol/L x 120 min). | 120 min
  Postprandial plasma GLP-1 area under the curve (mmol/L x 120 min).

SECONDARY OUTCOMES:
Postprandial plasma GIP area under the curve (mmol/L x 120 min) | 120 min
  Postprandial plasma GIP area under the curve (mmol/L x 120 min)
Postprandial plasma PYY area under the curve (mmol/L x 120 min) | 120 min
  Postprandial plasma PYY area under the curve (mmol/L x 120 min)
Subjective ratings of appetite (au) | 120 min
  Subjective ratings of appetite (au)

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Share anonymised data in publication form

REFERENCES:
- [Derived] Chen YC, Smith HA, Hengist A, Chrzanowski-Smith OJ, Mikkelsen UR, Carroll HA, Betts JA, Thompson D, Saunders J, Gonzalez JT. Co-ingestion of whey protein hydrolysate with milk minerals rich in calcium potently stimulates glucagon-like peptide-1 secretion: an RCT in healthy adults. Eur J Nutr. 2020 Sep;59(6):2449-2462. doi: 10.1007/s00394-019-02092-4. Epub 2019 Sep 17. PMID 31531707